CLINICAL TRIAL: NCT02939053
Title: Correlation of Bioimpedance Measurements From the SOZO Device With Pulmonary Arterial Pressure Measurements From the CardioMEMS HF System
Brief Title: Correlation of SOZO BIS Measures With CardioMEMS PA Pressure
Status: Completed | Type: Observational
Sponsor: ImpediMed Limited (Industry)
Collaborators: Baim Institute for Clinical Research (Other); Scripps Health (Other)
Responsible Party: Sponsor
Other Study IDs: IPD-SOZO-01
Record Dates: First submitted 2016-10-12; First posted 2016-10-19 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: NYHA Class III Heart Failure
Keywords: Bioimpedance spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Single-arm: All subjects enrolled will undergo measurements with the SOZO device daily for 30 days.
  Interventions: Device: SOZO

INTERVENTIONS:
Device: SOZO — The SOZO device is a bioimpedance spectroscopy device that measures bioimpedance parameters.

SUMMARY:
This study aims to establish the degree to which change in the ratio of ECF to TBW measured using the SOZO BIS device correlates with change in end-expiratory end-diastolic PAP measured using the CardioMEMS HF System (St. Jude Medical).

DETAILED DESCRIPTION:
This is a prospective, single-arm, observational, non-randomized clinical study that will enroll patients with heart failure who have had a CardioMEMS™ device implanted to monitor their diastolic pulmonary artery pressure. The study will recruit and enroll thirty participants. Participants will be monitored daily at home for a period of 30 days. Each day, the patient's diastolic pulmonary artery pressure will be measured by CardioMEMS™ and the ImpediMed's BIS technology. Participant's weight will also be taken each day.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. NYHA Class III HF.
3. Patient has undergone implantation of CardioMEMS HF System (St. Jude Medical).
4. Patient is characterized by at least one of the following:

   * CardioMEMS implanted within the previous 90 days
   * Received treatment with intravenous diuretics within the previous 30 days
   * Received dose escalation of oral diuretics at least twice within the previous 30 days
5. Patient is able to sit upright for BIS measurements.
6. Patient provides written informed consent and authorization to use and disclose health information.

Exclusion Criteria:

1. Patient is enrolled in a concurrent interventional study of an experimental treatment that may confound the results of this study, in the investigator's opinion.
2. Patient has a clinical condition that would not allow them to complete the study.
3. Patient is pregnant or lactating.
4. Patient has nephrotic syndrome or nephrosis.
5. Patient has estimated glomerular filtration rate (eGFR) < 20 ml/min/1.73m2 or end-stage renal disease requiring chronic dialysis.
6. Patient has been diagnosed with lymphedema.
7. Patient has chronic liver failure or cirrhosis.
8. Patient has a moderate or large pleural effusion as seen on chest X-ray.
9. Patient has been diagnosed with thrombophlebitis or deep vein thrombosis in arms or legs in the past 90 days.
10. Patient has an implanted cardiac rhythm management device (pacemaker or implantable cardioverter defibrillator).
11. Patient has an amputation of a limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients who have a cardioMEMS device
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Change in the ratio of whole body ECF/TBW measured using the SOZO BIS device | From baseline through study completion, an average of 30 days
  Changes of body fluid levels in heart failure patients

SECONDARY OUTCOMES:
Change in the ratio of thoracic ECF/TBW | From baseline through study completion, an average of 30 days
  Changes of thoracic fluid levels in heart failure patients
Change in the ratio of lower extremity ECF/TBW | From baseline through study completion, an average of 30 days
  Changes of lower limb fluid levels in heart failure patients

CONTACTS AND LOCATIONS:
Overall Officials: Roy Small, MD, Principal Investigator — Lancaster General Hospital
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Lancaster General Hospital, Lancaster, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
This is a pilot study, no individual participant data will be made available.

REFERENCES:
- [Derived] Accardi AJ, Matsubara BS, Gaw RL, Daleiden-Burns A, Heywood JT. Clinical Utility of Fluid Volume Assessment in Heart Failure Patients Using Bioimpedance Spectroscopy. Front Cardiovasc Med. 2021 Apr 7;8:636718. doi: 10.3389/fcvm.2021.636718. eCollection 2021. PMID 33898536